CLINICAL TRIAL: NCT01268735
Title: The Effect of Ocular Surface Lubricant Eyedrops on Lid Parallel Conjunctival Folds (LIPCOF) and Other Signs and Symptoms of Dysfunctional Tear Syndrome
Brief Title: The Effect of Ocular Lubricant Eyedrops on Lid Parallel Conjunctival Folds and Other Signs and Symptoms of Dry Eye
Acronym: LIPCOF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Igor Petricek, Ophthalmologist, Zagreb University Hospital Eye Department
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIPCOF Petricek
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Dry Eye Syndromes
Keywords: Dysfunctional Tear Syndrome; Dry Eye; LIPCOF; Hydroxypropyl-guar
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lubricating eyedrops containing HP-guar (Experimental)
  Interventions: Drug: Lubricating eyedrops containing hydroxypropyl-guar

INTERVENTIONS:
Drug: Lubricating eyedrops containing hydroxypropyl-guar — Eyedrops BID
  Other Names: Systane lubricating eyedrops, ALCON

SUMMARY:
Purpose To try to establish whether lid-parallel conjunctival folds (LIPCOF) can be influenced by increased lubrication with rewetting and lubricating eyedrops containing hydroxypropyl-guar, which has proven lubricating effect.

Methods During summer and fall of 2009, 16 ophthalmologists from various regions of Croatia investigated the effect of topical therapy with lubricating eyedrops on the signs and symptoms of dry eye, with the special emphasis on lid-parallel conjunctival folds (LIPCOF). 229 patients were enrolled in the study.

Results After 14 days of therapy with lubricating eyedrops containing hydroxypropyl-guar, statistically significant reduction of LIPCOF grade was observed, as well as the reduction of symptoms and other signs of dysfunctional tear syndrome (TBUT, Schirmer test, conjunctival hyperemia).

Conclusion Results of this study have shown positive influence of lubricating eyedrops containing hydroxypropyl-guar on signs and symptoms of dysfunctional tear syndrome even after only 14 days of treatment. It is of particular interest that LIPCOF grade was statistically significantly decreased, pointing at increased friction and decreased ocular surface lubrication as possible causes of its appearance.

Having this in mind, every clinician involved in dysfunctional tear syndrome treatment must also think about lubrication as integral part of treating this condition.

DETAILED DESCRIPTION:
Ruprecht et al. (1976-78) were among the first to ask a general population a simple question: "do you have gritty sensation in your eyes?". The results have shown that in the age group 55-59, 22,8% females and 9,9% males reported this symptom. In the age group 45-54 years, almost 20% of females and 15% of males also had dry eye signs. Based on reported symptoms, Schirmer test, TBUT test or Rose Bengal Staining, Jacobssson et al. in their survey among 780 subjects belonging to general population in Sweden have found that prevalence of dry eye in the age group 55-72 years was 15%. In the more recent study by Hikichi et al. in Japan, which screened 2127 patients in eight medical centers, dry eye symptoms were found among 17% of them. No seasonal fluctuations were observed. Survey on 504 subjects aged 30-60 in Kopenhagen has revealed the prevalence of dry eye in 11% of them. In a larger study in Maryland, USA, involving 2520 residents older than 65, 15% reported one or more dry eye symptoms, but only 2.2% of them also had pathological Schirmer test.

Mentioned studies have shown that dry eye symptoms were most prevalent in the age group older than 50, although no correlation was found between the age and gender. McCarthy et al. analyzed the prevalence of dry eye in Melbourne (Australia). 926 participants older than 40 were enrolled in the survey. Dry eye was diagnosed in 10.8% of subjects by Rose Bengal staining, in 16.3% of them by Schirmer test, 8.6% by TBUT test, 1.5% by fluorescein staining, in 7.4 of subjects by using two or more tests, and in 5.5% of subjects with the extreme symptoms of dry eye unrelated to hay fever. Women reported dry eye symptoms more frequently than men. Canadian Dry Eye Epidemiology Study (CANDEES) tried to establish the prevalence of dry eye in Canada. Questionnaires were mailed to every optometrist in Canada, who were asked to hand them out to 30 consecutive patients. The total of 13.517 completed questionnaires were returned (15.6% of those sent out). All age groups were enrolled in the study. 55% of subjects were in the age group 21-50, 60.7% were women, and 24.3% of them wore contact lenses. Dry eye symptoms were reported by 28.7% of surveyed subjects. When asked to describe the severity of symptoms, 7.6% reported moderate but constant symptoms, while 1.6% of them described them as severe. It is interesting to note that the vast majority of subjects who reported having severe symptoms were women (ratio women to men: 46:1). Regarding gender, 33% of women and 22% of men reported dry eye symptoms. Salisbury Study (1997) found dry eye symptoms in 59% of surveyed subjects. In Beaver Dam Eye Study (2000) 14,4% out of 3703 surveyed subjects had dry eye symptoms11. Part of this study was to analyze possible association of dry eye symptoms with other parameters. Statistically significant and independent association was found between dry eye symptoms and arthritis, smoking, coffee drinking, hyperthyreosis, goiter, diabetes and taking multivitamin food supplements.

When analyzing causes of first visits to the general outpatient office in Zagreb University Hospital Eye Department, 6.3% of all patients reported dysfunctional tear syndrome symptoms as their primary cause for visit. That percentage rose to 48% when only patients with external eye disease symptoms were analyzed, and would no doubt be even higher if only chronic external eye inflammatory conditions were counted.

Group of authors led by Prof.Hoeh 1995 published the paper Lid-parallel conjunctival folds are a sure diagnostic sign of dry eye. The method described was named Lidkantenparallelen Konjunktivalen Falten, or Lid Parallel Conjunctival Folds (LIPCOF). It was presented as a very useful and innovative way of diagnosing dry eye. However, it was up till now mentioned in relatively few published papers and is rarely used in everyday clinical practice, especially outside Europe, where it is frequently termed conjunctivochalasis and not associated with dry eye.

According to authors, the height and/or number of bulbar conjunctival folds parallel to the temporal margin of the lower eyelid are observed. Before assessment, lower eyelid is briefly lifted from the eye surface- if folds disappear, they indeed are what is described as LIPCOF.

Findings are ranked as follows:

Grade 0: no folds- normal finding (not dry eye) Grade 1: one fold above the normal tear meniscus height- mild dry eye Grade 2: multiple folds up to the height of normal tear meniscus- moderately dry eye Grade 3: multiple folds above normal tear meniscus height- severe dry eye Authors claim that LIPCOF has 93% positive predictive value. In other words, it detects dry eye with 93% certainty. Its negative predictive value is claimed to be 76%. Furthermore, LIPCOF is not invasive, takes very short time to perform and has no additional costs, as it requires use of no test strips, dyes etc.

Despite all mentioned advantages of this method, we still do not know what it actually measures- proven correlation between conjunctival folds and other signs and symptoms of dry eye does not automatically point at the reasons of their appearance.

One of the possible causes of LIPCOF may be decreased lubrication and increased friction of ocular surface and eyelids during blinking in dysfunctional tear syndrome. The importance of friction between the upper eyelid and ocular surface was well described by Korb in his Lid Wiper Epitheliopathy concept.

Nowadays, we have at our disposal commercially available rewetting eyedrops which, due to their formulation, display proven lubricating effect as well. If their application reduces LIPCOF grade, then increased friction may be the cause of the appearance of folds. Furthermore, such finding may show that this sign of dysfunctional tear syndrome may be influenced by appropriate therapy.

The aim of this study was to try to establish whether LIPCOF can be influenced by increased lubrication with rewetting and lubricating eyedrops containing hydroxypropyl-guar which has proven lubricating effect. Should that be the case, then it may be concluded that conjunctival folds appear due to the increased friction, and that they are dynamic condition, reversible after appropriate therapy. The influence of lubrication on other signs and symptoms of dry eye was also observed.

ELIGIBILITY:
Inclusion Criteria:

Ocular foreign body sensation, burning or stinging, complaints more pronounced in winter, windy conditions, during computer work, being bilateral, of the duration longer than three months, visual acuity fluctuations depending on blinking after longer reading or computer work, and tearing in cold weather, in the morning, after longer reading or computer work. Patients were also asked whether the symptoms were more pronounced in the morning or evening. The main enrollment criterion was the score of the above listed symptoms 15 or higher.

Exclusion Criteria:

Pregnant women, children, chronic eye patients on continuous topical therapy during previous month (i.e.glaucoma) and patients suffering from any acute eye disease and therefore on topical or systemic therapy in the previous month were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Lid-parallel conjunctival folds (LIPCOF) | 14 days
  The effect of topical therapy with lubricating eyedrops on lid-parallel conjunctival folds (LIPCOF).

SECONDARY OUTCOMES:
Signs and symptoms of dry eye | 14 days
  The effect of topical therapy with lubricating eyedrops on the signs and symptoms of dry eye.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Petricek, MD, Principal Investigator — Zagreb University Hospital Eye Department
Locations (1):
- Zagreb University Hospital Eye Department, Zagreb, Croatia